CLINICAL TRIAL: NCT06354842
Title: Application of Pilocarpine Iontophoresis in Patients With Chronic Kidney Disease: a Feasibility Study
Brief Title: Measurement of Sweat Sodium Concentration in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Tarik Shoumariyeh, Clinical resident & PhD student, Medical University of Vienna
Other Study IDs: 12345678
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Control: Healthy control subjects
  Interventions: Diagnostic Test: pilocarpine iontopheresis
- CKDI: Patients with chronic kidney disease G1
  Interventions: Diagnostic Test: pilocarpine iontopheresis
- CKDII: Patients with chronic kidney disease G2
  Interventions: Diagnostic Test: pilocarpine iontopheresis
- CKDIIIa: Patients with chronic kidney disease G3a
  Interventions: Diagnostic Test: pilocarpine iontopheresis
- CKDIIIb: Patients with chronic kidney disease G3b
  Interventions: Diagnostic Test: pilocarpine iontopheresis
- CKDIV: Patients with chronic kidney disease G4
  Interventions: Diagnostic Test: pilocarpine iontopheresis
- CKDV: Patients with chronic kidney disease G5
  Interventions: Diagnostic Test: pilocarpine iontopheresis
- CKDVd: Patients with chronic kidney disease G5 receiving hemodialysis
  Interventions: Diagnostic Test: pilocarpine iontopheresis

INTERVENTIONS:
Diagnostic Test: pilocarpine iontopheresis — Application of pilocarpine on the skin of the patients/subjects to induce sweat production to analyse sweat sodium concentration via flame photometry

SUMMARY:
It has been shown that excretion of sodium and water through the skin in the form of sweat represents a regulatory mechanism of electrolyte- and fluid balance. Since patients with chronic kidney disease (CKD) exhibit increased skin sodium content, we investigated the feasibility of sweat testing as a novel experimental tool to a more complete assessment of fluid- and sodium homeostasis.

In this cross-sectional feasibility study, we applied pilocarpine iontophoresis to induce sweat testing in 58 patients across various stages of CKD including patients after kidney transplantation as well as a healthy control cohort (n=6) to investigate possible effects of CKD and transplantation status on sweat rate and sodium concentration. Due to non-linear relationships, we modeled our data using polynomial regression.

Decline of kidney function showed a significant association with lower sweat rates: adj R²= 0.2278, F(2, 61) = 10.29, p = 0.000141. Sweat sodium concentrations were increased in moderate CKD, however this effect was lost in end stage renal disease: adj R² = 0.3701, F(4, 59) = 10.26, p = 2.261e-06. We observed higher sweat weight in males compared to females.

Diagnostic sweat analysis represents an innovative and promising noninvasive option for more thorough investigation of sodium- and fluid homeostasis in CKD patients. Lower sweat rates and higher sweat sodium concentrations represent a unique feature of CKD patients with potential therapeutic implications.

ELIGIBILITY:
Inclusion Criteria:

Completed 18th year of life and the ability and willingness to provide informed consent

Exclusion Criteria:

General exclusion criteria were signs of acute infection, clinical signs of kidney graft rejection or pregnancy. Exclusion criteria for the healthy controls were pregnancy or the presence of chronic metabolic, renal, cardiovascular, or rheumatologic conditions, hypertension, chronic or recent intake (8 weeks prior to testing) of psychiatric or antihypertensive medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls older than 18 years old. Patients older than 18 years old with all grades of Chronic Kidney Disease (also patients receiving hemodialysis)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Sweat sodium concentration | Right after study inclusion of patients/subjects
  Sodium concentration of induced sweat by pilocarpine iontopheresis in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Kovarik, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shoumariyeh T, Logar F, Helk O, Hofer J, Schmetterer KG, Mersi B, Gruber S, Saemann MD, Kaltenecker CC, Kovarik JJ. Decline of kidney function is associated with lower sweat weight in patients with chronic kidney disease. Sci Rep. 2025 Jul 2;15(1):22518. doi: 10.1038/s41598-025-05855-8. PMID 40596012